CLINICAL TRIAL: NCT01400152
Title: The Effect of Active Warming in Prehospital Trauma Care During Road and Air Ambulance Transportation - a Clinical Randomized Trial
Brief Title: Active Warming in Prehospital Trauma Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Ministry of Health and Social Affairs, Sweden (Other Government)
Responsible Party: Ulf Björnstig, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: jpl1
Record Dates: First submitted 2011-07-18; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Body Core Temperature; Thermal Comfort
Keywords: Hypothermia, body temperature regulation,thermal comfort, active warming, passive warming, prehospital trauma care
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Passive warming with additional active warming (Active Comparator)
  Interventions: Device: Additional active warming
- Passive warming (No Intervention)

INTERVENTIONS:
Device: Additional active warming — Chemical heat pad applied to the upper torso
  Arms: Passive warming with additional active warming

SUMMARY:
Prevention and treatment of hypothermia by active warming in prehospital trauma care is recommended but scientifical evidence of its effectiveness in a clinical setting is scarce. The objective of this study was to evaluate the effect of additional active warming during road or air ambulance transportation of trauma patients.

Patients were assigned to either passive warming with blankets or passive warming with blankets with the addition of an active warming intervention using a large chemical heat pad applied to the upper torso. Ear canal temperature, subjective sensation of cold discomfort and vital signs were monitored.

Mean core temperatures increased from 35.1°C (95% CI; 34.7-35.5 °C) to 36.0°C (95% CI; 35.7-36.3 °C) (p<0.05) in patients assigned to passive warming only (n=22) and from 35.6°C (95% CI; 35.2-36.0 °C) to 36.4°C (95% CI; 36.1-36.7°C) (p<0.05) in patients assigned to additional active warming (n=26) with no significant differences between the groups. Cold discomfort decreased in 2/3 of patients assigned to passive warming only and in all patients assigned to additional active warming, the difference in cold discomfort change being statistically significant (p<0.05). Patients assigned to additional active warming also presented a statistically significant decrease in heart rate and respiratory frequency (p<0.05).

In mildly hypothermic trauma patients, with preserved shivering capacity, adequate passive warming is an effective treatment to establish a slow rewarming rate and to reduce cold discomfort during prehospital transportation. However, the addition of active warming using a chemical heat pad applied to the torso will significantly improve thermal comfort even further and reduce the cold induced stress response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were sequential trauma patients, age ≥ 18 years, who had sustained an injury outdoors and were transported by one of the participating EMS units.

Exclusion Criteria:

* Patients were excluded if initial level of consciousness was affected, (Glasgow Coma Scale < 15), if they required prehospital CPR or if duration of transportation was expected to be shorter than 10 minutes.
* As the aim of the study was to investigate the effect of active warming intervention in cold stressed patients, those patients who had already received active warming or had been taken indoors for more than 10 minutes before EMS unit arrival or had an initial cold discomfort rating ≤ 2 were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Body core temperature | From initial assessment upon arrival of EMS crew until second assessment about 30 minutes later.
Cold discomfort | From initial assessment upon arrival of EMS crew until second assessment about 30 minutes later.

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Björnstig, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Department of Surgery and Perioperative Sciences, Umeå University, Umeå, Sweden

REFERENCES:
- [Derived] Lundgren P, Henriksson O, Naredi P, Bjornstig U. The effect of active warming in prehospital trauma care during road and air ambulance transportation - a clinical randomized trial. Scand J Trauma Resusc Emerg Med. 2011 Oct 21;19:59. doi: 10.1186/1757-7241-19-59. PMID 22017799